CLINICAL TRIAL: NCT04050943
Title: A Long-term, Prospective, Observational Cohort of Patients With Chronic Pulmonary Disease
Brief Title: A Cohort of Patients With Chronic Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guan Lili, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GIRH-CRD2019
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRD patients: Patients with chronic pulmonary disease like COPD, asthma, bronchiectasis, and etc.
  Interventions: Other: observational cohort

INTERVENTIONS:
Other: observational cohort — Recording the clinical, pathophysiology, and psychological parameters, to observe and predict the clinical outcomes of these patients.

SUMMARY:
This is a longitudinal study of following chronic pulmonary disease patients to observe and predict the clinical outcomes of these patients.

DETAILED DESCRIPTION:
In patients with chronic pulmonary disease, impaired pulmonary function and limited exercise capacity, is a complex clinical syndrome with a wide range of underlying causes, which may result in worse quality of life and high economic burden. This is a longitudinal study of following chronic pulmonary disease patients, recording the clinical, pathophysiology, and psychological parameters, to observe and predict the clinical outcomes of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80, males and females
2. Patients are diagnosed as the obstructive pulmonary disease according to the clinical practice.
3. Willing to participate in the study.
4. Being able to provide informed consent.

Exclusion Criteria:

1. Subjects with severe heart failure, severe arrhythmias, unstable angina, and malignant comorbidities.
2. Subjects with significantly impaired cognitive function and are unable to fulfill the study requirement (unable to provide informed consent)
3. Subjects who participated in another trial within 30 days prior to the planned start of the study
4. Subjects with cancer or have had cancer in the 5 years prior to study entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a longitudinal study of following obstructive pulmonary disease patients from the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of acute exacerbations | 1 year
  The rate of exacerbations within 1 year of these patients will be tracked.

SECONDARY OUTCOMES:
Survival | 1 year
  The rate of survival within 1 year of these patients will be tracked.
Forced expiratory volume in 1 second | 1 year
  Forced expiratory volume in 1 second is a marker used to measure lung function and can help you monitor your lung diseases over time.
Health related quality of life: questionnaires | 1 year
  Using questionnaires to reflect the patients' health related quality of life.
  The questionnaires include:
  1. SF-36 (scores range between 0 and 100 and higher scores are attributed to better quality of life.)
  2. St. George's Respiratory Questionnaire (scores range between 0 and 100 and higher scores are attributed to worse quality of life.)
  3. Severe Respiratory Insufficiency Questionnaire (scores range between 0 and 100 and higher scores are attributed to better quality of life.)
6-minute walk test | 1 year
  The 6-minute walk test plays a key role in evaluating functional exercise capacity, assessing prognosis and evaluating response to treatment across a wide range of respiratory diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China